CLINICAL TRIAL: NCT03927963
Title: The Anti-inflammatory Effect and Hemodynamic Stability of Dexmedetomidine in Aneurysmal Clipping Operation; Compare With Propofol
Brief Title: The Neuroprotection Effect of Dexmedetomidine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Jiyoung Yoo, Assistant professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: AJIRB-MED-OBS-18-478
Record Dates: First submitted 2019-03-12; First posted 2019-04-25 (Actual); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Dexmedetomidine
MeSH Terms: interventions — Dexmedetomidine; Propofol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- propofol (Placebo Comparator)
  Interventions: Drug: Propofol
- dexmedetomidine (Active Comparator)
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine 0.7 ug/kg/h with sevoflurane 0.5 MAC and remifentanil infusion are used throughout anesthesia period
  Arms: dexmedetomidine
Drug: Propofol — Effect site concentration of propofol 1.5 ng/ml with sevoflurane 0.5 MAC and remifentanil infusion are used throughout anesthesia period
  Arms: propofol

SUMMARY:
The brain protection effect of dexmedetomidine has been approved in several studies.

Basically, the anti-inflammatory effects and reducing catecholamines are thought to be a main role of the protection effect. In many studies reported the advantage of dexmedetomidine as a substitution of other sedative drugs for anesthesia.

The anesthesia of intra-cranial aneurysmal clipping operation commonly use intravenous anesthetic agents combined with inhalation anesthesia for neuroprotection, and mostly propofol is used.

The aim of this study is to examine the effects of dexmedetomidine on serum inflammatory markers and research the hemodynamic stability of dexmedetomidine compared to propofol in aneurysmal clipping operation.

ELIGIBILITY:
Inclusion Criteria:

* ASA class I,II patient needs operation of intracranial aneurysmal clipping without SAH

Exclusion Criteria:

* Any history of neurologic disease, dementia
* Allergic history of propofol or dexmedetomidine

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2019-05-01 (Estimated); Primary Completion 2020-09-30 (Estimated); Study Completion 2021-02-28 (Estimated)

PRIMARY OUTCOMES:
The concentration of inflammatory markers | Baseline: Before injection study drugs
  CRP (mg/ml)
The concentration of inflammatory markers | 1 minute after operation
  CRP (mg/ml)
The concentration of inflammatory markers | Day 1 after operation
  CRP (mg/ml)
The concentration of inflammatory markers | Day 2 after operation
  CRP (mg/ml)
The concentration of norepinephrine | Baseline: Before injection study drugs
  NE (nmol/l)
The concentration of norepinephrine | 1 minute after operation
  NE (nmol/l)
The concentration of norepinephrine | Day 1 after operation
  NE (nmol/l)
The concentration of norepinephrine | Day 2 after operation
  NE (nmol/l)
The concentration of inflammatory markers | Baseline: Before injection study drugs
  IL-6, IL-8, IL-10 ,TNF-a (pg/ml)
The concentration of inflammatory markers | 1 minute after operation
  IL-6, IL-8, IL-10 ,TNF-a (pg/ml)
The concentration of inflammatory markers | Day 1 after operation
  IL-6, IL-8, IL-10 ,TNF-a (pg/ml)
The concentration of inflammatory markers | Day 2 after operation
  IL-6, IL-8, IL-10 ,TNF-a (pg/ml)

SECONDARY OUTCOMES:
The frequency of hypotension or hypertension | during operation

IPD SHARING:
Plan to Share IPD: Undecided